CLINICAL TRIAL: NCT01986062
Title: A Multicenter, Dose-Optimized, Double-Blind, Randomized, Placebo-Controlled, Crossover Study to Evaluate the Efficacy of AR11 (Amphetamine Sulfate) in Pediatric Patients (Ages 6-12) With ADHD in a Laboratory Classroom
Brief Title: Crossover Study to Evaluate the Efficacy of AR11 in Pediatric Patients With ADHD in a Laboratory Classroom Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR11.001
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Results first posted 2016-04-19 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2016-03

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; AR11; classroom design; amphetamine sulfate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AR11 (amphetamine sulfate) (1 week) - double blind (Experimental): AR11, administered orally, BID, for one week (crossover to placebo administration week 2)
  Interventions: Drug: AR11
- Placebo (1 week) - double blind (Placebo Comparator): Placebo, administered orally, BID, for one week (crossover to AR11 administration week 2)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AR11
  Other Names: amphetamine sulfate
  Arms: AR11 (amphetamine sulfate) (1 week) - double blind
Drug: Placebo
  Other Names: matching Placebo
  Arms: Placebo (1 week) - double blind

SUMMARY:
This is a dose-optimized, randomized, double-blind, placebo-controlled crossover study in approximately 100 pediatric patients (aged 6 to 12 years) with ADHD. Eligible patients will enroll to take open-label AR11 BID and undergo dose optimization activities for 8 weeks. Patients who achieve a stable dose during the dose optimization period will continue participation and will be randomized to take double-blind medication (AR11 or placebo) orally twice daily for 1 week. At the end of each double-blind treatment period, patients will be evaluated for ADHD symptoms in a laboratory classroom setting utilizing SKAMP and PERMP assessments.

DETAILED DESCRIPTION:
This is a dose-optimized, randomized, double-blind, placebo-controlled crossover study in approximately 100 pediatric patients (aged 6 to 12 years) with ADHD. Eligible patients will enroll in the study to take open-label AR11 twice daily and undergo dose optimization activities for 8 weeks. Patients who achieve a stable dose during the dose optimization period will continue participation and will be randomized to take double-blind medication (AR11 or placebo) orally twice daily for 1 week. At the end of the first double-blind treatment period, patients will be evaluated for ADHD symptoms in a laboratory classroom setting utilizing SKAMP and PERMP assessments. At the end of the second double blind treatment period, patients will be evaluated for ADHD symptoms in a second laboratory classroom setting utilizing SKAMP and PERMP assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 6 and 12 years of age, inclusive, at the time of Screening.
2. Diagnosed as meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for ADHD.
3. A clinician-administered Clinical Global Impression of Severity (CGI-S) score of 3 or greater.
4. An ADHD Rating Scale (ADHD-RS) score at Screening and Baseline greater than or equal to the 90th percentile normative values for gender and age in at least one of the following categories: hyperactive-impulsive subscale, inattentive subscale, or total score.

Exclusion Criteria:

1. Secondary or co-morbid diagnoses other than ADHD, with the exception of simple phobias, oppositional defiant disorder, elimination disorders, motor skills disorders, communication disorders, learning disorders, adjustment disorders, and sleep disorders if, in the opinion of the investigator, the associated symptoms do not confound assessment of safety or efficacy.
2. Clinically significant cognitive impairment as assessed in the clinical judgment of the Investigator.
3. History of any of the following medical disorders: seizure disorder (excluding a history of febrile seizures), structural cardiac disorders, serious cardiac conditions, hypertension, untreated thyroid disease, glaucoma, Tourette's disorder, or chronic tics.
4. Clinically significant abnormal ECG finding or abnormal cardiac finding on physical exam (including presence of a pathologic murmur) at Screening.
5. Use of any psychotropic medication (sedative hypnotics prescribed as a sleep aid at a stable dose for at least 30 days prior to Baseline, at bedtime only, are allowed during the study).
6. A history of hypersensitivity or intolerance to any formulation of amphetamine or lisdexamfetamine.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Downey, MD, Study Director — Arbor Pharmaceuticals, LLC.
Locations (7):
- United States (7):
  - Florida Clinical Research Center, LLC., Bradenton, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Miami Research Associates, South Miami, Florida
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Duke University Medical Center, Durham, North Carolina
  - Bayou City Research Ltd., Houston, Texas
  - Westex Clinical Investigations, Houston, Texas

REFERENCES:
- [Background] Childress AC, Brams M, Cutler AJ, Kollins SH, Northcutt J, Padilla A, Turnbow JM. The Efficacy and Safety of Evekeo, Racemic Amphetamine Sulfate, for Treatment of Attention-Deficit/Hyperactivity Disorder Symptoms: A Multicenter, Dose-Optimized, Double-Blind, Randomized, Placebo-Controlled Crossover Laboratory Classroom Study. J Child Adolesc Psychopharmacol. 2015 Jun;25(5):402-14. doi: 10.1089/cap.2014.0176. Epub 2015 Feb 18. PMID 25692608
- [Derived] Childress AC, Newcorn JH, Cutler AJ. Gender Effects in the Efficacy of Racemic Amphetamine Sulfate in Children with Attention-Deficit/Hyperactivity Disorder. Adv Ther. 2019 Jun;36(6):1370-1387. doi: 10.1007/s12325-019-00942-5. Epub 2019 Apr 10. PMID 30972657

RESULTS

PARTICIPANT FLOW:
Groups:
- AR11 (1 Week) Then Placebo (1 Week) - Double Blind: AR11, administered orally, BID, for one week (crossover to placebo administration week 2)
- Placebo (1 Week) Then AR11 (1 Week) - Double Blind: Placebo, administered orally, BID, for one week (crossover to AR11administration week 2)
Period: Overall Study
Arm/Group | AR11 (1 Week) Then Placebo (1 Week) - Double Blind | Placebo (1 Week) Then AR11 (1 Week) - Double Blind
Started | 47 | 50
Completed | 46 | 49
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- AR11 (1 Week) Then Placebo (1 Week) - Double Blind: AR11, administered orally, BID for one week (crossover to placebo administration week 2)
- Placebo (1 Week) Then AR11 (1 Week) - Double Blind: Placebo, administered orally, BID for one week (crossover to AR11 administration week 2)
- Total: Total of all reporting groups
Arm/Group | AR11 (1 Week) Then Placebo (1 Week) - Double Blind | Placebo (1 Week) Then AR11 (1 Week) - Double Blind | Total
Number analyzed (Participants) | 47 | 50 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.6 (1.97) | 9.6 (1.78) | 9.6 (1.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 29 | 30 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 20 | 33
  White | 30 | 28 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 47 | 50 | 97

OUTCOME MEASURES:

1. Primary Outcome: SKAMP-Combined Scores
Description: Swanson, Kotkin, Agler, M-Flynn, and Pelham Scale [SKAMP]-combined scores measured during Laboratory Classroom Days. The SKAMP scale is a validated subjective measure of ADHD symptoms in a laboratory classroom, comprised of 13 items on which subjects are rated according to a 7 point scale (0=normal to 6=maximal impairment); maximum score 78. The SKAMP-combined score is obtained by summing the rating values for each of the 13 items, whereby the higher the SKAMP score, the greater the impairment.
Time Frame: 2 hours post-dose
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- AR11 (Amphetamine Sulfate): AR11, administered orally, BID, 10-40 mg/day
- Placebo: Placebo, administered orally, BID
Arm/Group | AR11 (Amphetamine Sulfate) | Placebo
Number analyzed (Participants) | 95 | 97
units on a scale | 10.0 (8.24) | 17.8 (1.94)
Statistical Analysis 1: Comparison: AR11 (Amphetamine Sulfate) vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

2. Secondary Outcome: SKAMP-Combined Scores
Description: as for outcome 1
Time Frame: 0.75, 4, 6, 8, 10 hours post-dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AR11 (Amphetamine Sulfate) | Placebo
Number analyzed (Participants) | 95 | 97
units on a scale
  0.75 hours post-dose | 11.8 (10.56) | 17.3 (11.38)
  4 hours post-dose | 11.6 (10.04) | 19.8 (11.92)
  6 hours post-dose | 14.5 (10.38) | 20.2 (11.28)
  8 hours post-dose | 16.0 (11.76) | 22.0 (12.33)
  10 hours post-dose | 16.5 (11.08) | 20.8 (13.33)
Statistical Analysis 1: Comparison: AR11 (Amphetamine Sulfate) vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

3. Secondary Outcome: SKAMP Subscale - Attention Scores
Description: The SKAMP scale is a validated subjective measure of ADHD symptoms. It is comprised of 13 items (grouped under the subcategories of attention, deportment, quality of work, and compliance) on which subjects are rated according to a 7-point scale (0 = normal to 6 = maximal impairment). The SKAMP-Attention subscale score is comprised of four of the 13 items with a maximum score of 24.
Time Frame: 0.75, 2, 4, 6, 8, and 10 hours post-dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AR11 (Amphetamine Sulfate) | Placebo
Number analyzed (Participants) | 95 | 97
units on a scale
  0.75 hours post-dose | 2.2 (2.64) | 3.4 (3.06)
  2.0 hours post-dose | 1.9 (2.26) | 3.4 (3.1)
  4.0 hours post-dose | 2.2 (2.68) | 4.0 (3.04)
  6.0 hours post-dose | 2.3 (2.43) | 3.6 (2.95)
  8.0 hours post-dose | 2.8 (2.8) | 4.1 (3.01)
  10.0 hours post-dose | 3.2 (3.15) | 4.0 (3.59)
Statistical Analysis 1: Comparison: AR11 (Amphetamine Sulfate) vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

4. Secondary Outcome: SKAMP Subscale - Deportment Scores
Description: The SKAMP scale is a validated subjective measure of ADHD symptoms. It is comprised of 13 items (grouped under the subcategories of attention, deportment, quality of work, and compliance) on which subjects are rated according to a 7-point scale (0 = normal to 6 = maximal impairment). The SKAMP-Deportment subscale score is comprised of four of the 13 items with a maximum score of 24.
Time Frame: 0.75, 2, 4, 6, 8, and 10 hours post-dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AR11 (Amphetamine Sulfate) | Placebo
Number analyzed (Participants) | 95 | 97
units on a scale
  0.75 hours post-dose | 2.1 (3.53) | 3.9 (4.82)
  2.0 hours post-dose | 1.6 (2.79) | 4.0 (4.58)
  4.0 hours post-dose | 2.1 (3.47) | 4.7 (4.86)
  6.0 hours post-dose | 3.1 (4.21) | 4.3 (4.51)
  8.0 hours post-dose | 3.5 (4.38) | 4.9 (4.8)
  10.0 hours post-dose | 3.1 (3.72) | 4.9 (5.21)
Statistical Analysis 1: Comparison: AR11 (Amphetamine Sulfate) vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

5. Secondary Outcome: PERM-P Scores - Number of Problems Attempted
Description: Permanent Product Measure of Performance (PERMP) assessments measured during Laboratory Classroom Days. The PERMP is an individualized, five-page math exam consisting of 400 problems. Subjects are instructed to complete as many math problems as possible in 10 minutes. Performance is evaluated using the number of problems attempted (maximum score = 400) and the number of problems correct (maximum score = 400).
Time Frame: 0.75, 2, 4, 6, 8, and 10 hours post-dose
Population: ITT
Measure: Mean (Standard Deviation); unit: number of problems attempted
Arm/Group | AR11 (Amphetamine Sulfate) | Placebo
Number analyzed (Participants) | 95 | 97
number of problems attempted
  0.75 hours post-dose | 111.6 (53.53) | 91.2 (47.35)
  2.0 hours post-dose | 113.4 (51.27) | 85.7 (46.66)
  4.0 hours post-dose | 113.2 (56.28) | 85.1 (45.89)
  6.0 hours post-dose | 101.3 (54.26) | 74.9 (43.08)
  8.0 hours post-dose | 98.2 (56.11) | 76.4 (47.74)
  10.0 hours post-dose | 95.2 (55.53) | 76.3 (45.27)
Statistical Analysis 1: Comparison: AR11 (Amphetamine Sulfate) vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

6. Secondary Outcome: PERM-P Scores - Number of Problems Correct
Description: as for outcome 5
Time Frame: 0.75, 2, 4, 6, 8, and 10 hours post-dose
Population: ITT
Measure: Mean (Standard Deviation); unit: number of problems correct
Arm/Group | AR11 (Amphetamine Sulfate) | Placebo
Number analyzed (Participants) | 95 | 97
number of problems correct
  0.75 hours post-dose | 104.5 (54.49) | 83.9 (46.96)
  2.0 hours post-dose | 107.1 (53.15) | 78.9 (44.62)
  4.0 hours post-dose | 107.0 (57.46) | 79.9 (45.56)
  6.0 hours post-dose | 95.6 (55.43) | 70.5 (43.23)
  8.0 hours post-dose | 92.7 (57.28) | 71.5 (47.43)
  10.0 hours post-dose | 89.9 (55.29) | 72.3 (45.19)
Statistical Analysis 1: Comparison: AR11 (Amphetamine Sulfate) vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: AE reporting occurred during the 8-week open label treatment phase (i.e. AR11 dose optimization) and the 2-week double blind phase (i.e. crossover period)
Groups:
- AR11: AR11, administered orally, BID for one week
- Placebo: Placebo, administered orally, BID for one week
Arm/Group | AR11 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/97
Other Adverse Events (participants affected / at risk) | 19/97 | 6/97
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AR11 (N=97) | Placebo (N=97)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Mood swings (Psychiatric disorders) | 2 (2) | 0 (0)
Upper abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 3 (3)
Decreased weight (Investigations) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less